CLINICAL TRIAL: NCT02840487
Title: VRC 319: A Phase I/Ib, Randomized Clinical Trial to Evaluate the Safety and Immunogenicity of A Zika Virus DNA Vaccine, VRC-ZKADNA085-00-VP, in Healthy Adults
Brief Title: Safety and Immunogenicity of a Zika Virus DNA Vaccine, VRC-ZKADNA085-00-VP, in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 160148; 16-I-0148
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03-14

CONDITIONS: Prevention of Zika Infection; Zika-Specific Immune Response
Keywords: Zika Infection; Flavivirus; Vaccine-Mediated Protection; Immune Response; Arthropod-Borne Virus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (4):
- Group 1 (Experimental): ZIKV DNA vaccine administered IM at a dosage of 4mg, as two 0.5ml injections on Day 0 and Week 8.
  Interventions: Biological: VRC-ZKADNA085-00-VP
- Group 2 (Experimental): ZIKV DNA vaccine administered IM at a dosage of 4mg, as two 0.5ml injections on Day 0 and Week 12.
  Interventions: Biological: VRC-ZKADNA085-00-VP
- Group 3 (Experimental): ZIKV DNA vaccine administered IM at a dosage of 4mg, as two 0.5ml injections on Day 0, Week 4 and Week 8.
  Interventions: Biological: VRC-ZKADNA085-00-VP
- Group 4 (Experimental): ZIKV DNA vaccine administered IM at a dosage of 4mg, as two 0.5ml injections on Day 0,Week 4 and Week 20.
  Interventions: Biological: VRC-ZKADNA085-00-VP

INTERVENTIONS:
Biological: VRC-ZKADNA085-00-VP — VRC-ZKADNA085-00-VP is an investigational ZIKV DNA vaccine that is intended to prevent Zika virus infection.

SUMMARY:
Background:

The Zika virus is passed to humans by infected mosquitos. It usually causes fever, rash, joint pain, and red eyes. Recently, some cases of microcephaly (abnormally small head) were reported in babies born to mothers infected with the Zika virus. Rare cases of a severe nerve weakness called Guillain-Barr(SqrRoot)(Copyright) syndrome were reported in some people with Zika virus infection. There is currently no cure for or vaccine against the infection. VRC-ZKADNA085-00-VP is a new vaccine that instructs the body to make a small amount of Zika virus protein. The body may use this to build an immune response.

Objective:

To see if VRC-ZKADNA085-00-VP is safe and causes any side effects.

Eligibility:

Healthy people ages 18 35

Design:

Participants will be screened through a separate protocol with:

* Medical history
* Physical exam
* Lab and urine tests

Participants will be randomly assigned to 1 of 4 study groups. They will have about 18 clinic visits over 2 years. Most will occur in the first year, with long-term follow-up visits at months 18 and 24. Visits include a physical exam and blood and urine tests.

Participants will have vaccine injections. A high-pressure device pushes the vaccine through the skin and into the muscle of the upper arm. They will have 2-3 injections depending on their group.

Vaccine visits last 4-6 hours. Others last 1-2 hours.

Participants will keep a diary for 7 days after each injection. They will record their temperature and measure any skin changes at the injection site each day.

Participants might have extra visits and blood tests if they have health changes.

DETAILED DESCRIPTION:
Study Design:

This is a Phase I/Ib, randomized, multicenter clinical study to evaluate the safety, tolerability, and immunogenicity of four vaccination regimens against Zika virus (ZIKV) disease. Vaccination regimens with the VRC-ZKADNA085-00-VP (ZIKV DNA) vaccine administered on Day 0 and Week 8 (Group 1); on Day 0 and Week 12 (Group 2); on Day 0, Weeks 4 and 8 (Group 3); and on Day 0, Weeks 4 and 20 (Group 4) will be tested. The primary hypothesis is that the ZIKV DNA vaccine will be safe and well tolerated in healthy adults. A secondary hypothesis is that all vaccine regimens will elicit a ZIKV-specific immune response. The primary objectives are to evaluate the safety and tolerability of the investigational vaccine regimens in healthy adults. Secondary objectives are related to the immunogenicity of the vaccination regimens.

Product Description:

The investigational VRC-ZKADNA085-00-VP vaccine was developed by the Vaccine Research Center (VRC), NIAID, and is composed of a single closed-circular DNA plasmid that encodes the wild type precursor transmembrane M (prM) and envelope (E) proteins from the H/PF/2013 strain of ZIKV. Vaccine is supplied in single dose vials at a concentration of 4 mg/mL. ZIKV DNA vaccine dose will be 4 mg administered as an intramuscular (IM) injection in the deltoid muscle.

Subjects:

Healthy adults 18 to 35 years of age.

Study Plan:

Subjects will be enrolled at up to 3 study sites, randomized equally into the 4 study groups, and will receive 2-3 vaccinations. The protocol requires up to 18 scheduled clinic visits and a telephone follow-up contact after each study injection. Solicited reactogenicity will be evaluated using a 7-day diary card. Assessment of vaccine safety will include clinical observation and monitoring of hematological and chemical parameters at clinical visits through the 44 weeks on the study.

-VRC 319 Study Schema

* Group:1; Subjects*: 20; Day 0; Week 8;
* Group:2; Subjects*: 20; Day 0; Week 12;
* Group:3; Subjects*: 20; Day 0; Week 4; Week 8;
* Group:4; Subjects*: 20; Day 0; Week 4; Week 20;
* TOTAL; Subjects*: 80

  * Up to 120 total enrollments are permitted if additional subjects are needed for assessment of safety and immune responses.

Study Duration:

Subjects will be evaluated for safety and immune responses throughout the study for 44 weeks following the first vaccine administration and for durability of immune responses at two additional long term follow-up visits at 18 and 24 months.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18 to 35 years old
  2. Available for clinic visits for 24 months after enrollment
  3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
  4. Able and willing to complete the informed consent process
  5. Willing to donate blood for sample storage to be used for future research
  6. In good general health without clinically significant medical history
  7. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than or equal to 40 within the 56 days prior to enrollment
  8. Agrees not to receive licensed or investigational flavivirus vaccines through 4 weeks after last study injection

     INCLUSION CRITERIA - LABORATORY CRITERIA WITHIN 56 DAYS PRIOR TO ENROLLMENT:
  9. Hemoglobin within institutional normal limits or accompanied by the site PI or designee approval
  10. WBC and differential either within institutional normal range or accompanied by site PI or designee approval
  11. Total lymphocyte count greater than or equal to 800 cells/mm^3
  12. Platelets = 125,000 - 500,000/mm^3
  13. Alanine aminotransferase (ALT) less than or equal to 1.25 x institutional upper limit of normal (ULN)
  14. Serum creatinine less than or equal to 1.1 x institutional ULN
  15. Negative for HIV infection by an FDA approved method of detection

      INCLUSION CRITERIA - CRITERIA APPLICABLE TO WOMEN OF CHILDBEARING POTENTIAL:
  16. Negative human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) on day of enrollment
  17. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through 12 weeks after the last study vaccination

EXCLUSION CRITERIA - FEMALE-SPECIFIC:

1. Breast-feeding or planning to become pregnant while participating through 12 weeks after the last study vaccination

   EXCLUSION CRITERIA - SUBJECT HAS RECEIVED ANY OF THE FOLLOWING:
2. More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
3. Blood products within 16 weeks prior to enrollment
4. Inactivated vaccines within 2 weeks prior to enrollment
5. Live attenuated vaccines within 4 weeks prior to enrollment
6. Investigational research products within 4 weeks prior to enrollment or planning to receive investigational products while on the study
7. Current allergen immunotherapy with antigen injections, unless on maintenance schedule
8. Current anti-TB prophylaxis or therapy

   EXCLUSION CRITERIA - SUBJECT HAS A HISTORY OF ANY OF THE FOLLOWING CLINICALLY SIGNIFICANT CONDITIONS:
9. Laboratory confirmed ZIKV infection by self-report
10. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the site investigator
11. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
12. Asthma that is not well controlled
13. Diabetes mellitus (type I or II), with the exception of gestational diabetes
14. Evidence of autoimmune disease or immunodeficiency
15. Idiopathic urticaria within the past year
16. Hypertension that is not well controlled
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
18. Malignancy that is active or history of malignancy that is likely to recur during the period of the study
19. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
20. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
21. Guillain-Barre Syndrome, Bell s palsy or similar neurological conditions
22. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within 5 years prior to enrollment, a history of suicide plan or attempt
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-08-02; Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of four vaccination regimens with ZIKV DNA vaccine (VRC-ZKADNA085-00-VP) administered IM at 4 mg. | Through 44 weeks of study participation

SECONDARY OUTCOMES:
To evaluate the magnitude and frequency of ZIKV-specific antibodyresponse as measured by neutralization assay. | Four weeks after the second and third injections for each regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Gaudinski, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (3):
  - Hope Clinic - Emory Vaccine Ctr, Decatur, Georgia
  - University of Maryland Ctr. for Vaccine Development, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Background] Fauci AS, Morens DM. Zika Virus in the Americas--Yet Another Arbovirus Threat. N Engl J Med. 2016 Feb 18;374(7):601-4. doi: 10.1056/NEJMp1600297. Epub 2016 Jan 13. No abstract available. PMID 26761185
- [Background] Ledgerwood JE, Pierson TC, Hubka SA, Desai N, Rucker S, Gordon IJ, Enama ME, Nelson S, Nason M, Gu W, Bundrant N, Koup RA, Bailer RT, Mascola JR, Nabel GJ, Graham BS; VRC 303 Study Team. A West Nile virus DNA vaccine utilizing a modified promoter induces neutralizing antibody in younger and older healthy adults in a phase I clinical trial. J Infect Dis. 2011 May 15;203(10):1396-404. doi: 10.1093/infdis/jir054. Epub 2011 Mar 11. PMID 21398392
- [Background] Chang LJ, Dowd KA, Mendoza FH, Saunders JG, Sitar S, Plummer SH, Yamshchikov G, Sarwar UN, Hu Z, Enama ME, Bailer RT, Koup RA, Schwartz RM, Akahata W, Nabel GJ, Mascola JR, Pierson TC, Graham BS, Ledgerwood JE; VRC 311 Study Team. Safety and tolerability of chikungunya virus-like particle vaccine in healthy adults: a phase 1 dose-escalation trial. Lancet. 2014 Dec 6;384(9959):2046-52. doi: 10.1016/S0140-6736(14)61185-5. Epub 2014 Aug 14. PMID 25132507
- [Derived] Gaudinski MR, Houser KV, Morabito KM, Hu Z, Yamshchikov G, Rothwell RS, Berkowitz N, Mendoza F, Saunders JG, Novik L, Hendel CS, Holman LA, Gordon IJ, Cox JH, Edupuganti S, McArthur MA, Rouphael NG, Lyke KE, Cummings GE, Sitar S, Bailer RT, Foreman BM, Burgomaster K, Pelc RS, Gordon DN, DeMaso CR, Dowd KA, Laurencot C, Schwartz RM, Mascola JR, Graham BS, Pierson TC, Ledgerwood JE, Chen GL; VRC 319; VRC 320 study teams. Safety, tolerability, and immunogenicity of two Zika virus DNA vaccine candidates in healthy adults: randomised, open-label, phase 1 clinical trials. Lancet. 2018 Feb 10;391(10120):552-562. doi: 10.1016/S0140-6736(17)33105-7. Epub 2017 Dec 5. PMID 29217376